CLINICAL TRIAL: NCT01438853
Title: The Safety, Pharmacokinetics, and Pharmacodynamic Effects of TNX-832 (Sunol cH36) in Subjects With Acute Lung Injury/Acute Respiratory Distress Syndrome
Brief Title: Effects of TNX-832 (Sunol cH36) in Subjects With Acute Lung Injury/Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Collaborators: Genentech, Inc. (Industry); Tanox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNX-832.201
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Sepsis; Acute Lung Injury; Acute Respiratory Distress Syndrome; ALI/ARDS; Lung Disease
MeSH Terms: conditions — Sepsis; Acute Lung Injury; Respiratory Distress Syndrome; Lung Diseases | interventions — ALT-836

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNX-832 (Experimental): Anti-tissue factor antibody
  Interventions: Biological: TNX-832
- Drug Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: TNX-832 — Single intravenous dose of TNX-832 at 0.06, 0.08 or 0.10 mg/kg
  Other Names: ALT-836; Sunol cH36
  Arms: TNX-832
Drug: Placebo — Single intravenous dose of saline control
  Arms: Drug Placebo

SUMMARY:
This Phase I/IIa, multi-center, randomized, placebo-controlled, single-blinded dose-escalation study evaluated TNX-832 (also referred to as ALT-836 and Sunol cH36) in subjects with suspected or proven bacteria-induced ALI/ARDS. Up to five cohorts of at least six subjects each were originally planned. Subjects were to be randomized in a 5:1 ratio to receive TNX-832 or placebo,respectively, administered as a single bolus infusion over 15 minutes. Three cohorts of subjects were enrolled to the study and safety and pharmacokinetics of the study treatment were evaluated.

DETAILED DESCRIPTION:
Tissue factor (TF) is a transmembrane glycoprotein that acts as the principal initiator of the extrinsic coagulation pathway. TF is a key mediator between the immune system and coagulation and is the principal activator of coagulation. The TF-FVIIa complex activates FX and FIX, resulting in the cleavage of prothrombin to thrombin. Normally, localized activation of the coagulation cascade associated with inflammatory responses plays a role in controlling the spread of infectious agents; however, aberrant TF expression often leads to serious thrombotic disorders. TF-dependent thrombosis has been associated with many diseases including septic shock, coronary artery disease (CAD), cancer, and many inflammatory and autoimmune disorders such as lupus, rheumatoid arthritis, psoriasis, and inflammatory bowel disease.

Acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are forms of acute respiratory failure characterized by diffuse pulmonary infiltrates, pulmonary hypertension, refractory hypoxemia, loss of pulmonary compliance and normal hydrostatic pressures. ALI and ARDS commonly occur in patients with acute catastrophic events such as sepsis, trauma and severe pulmonary infections. The incidence of ALI and ARDS is extremely high in patients with sepsis. By blocking the initiating events of extrinsic coagulation activation, their effects on pro-inflammatory events in the lungs and disordered fibrin deposition may be corrected and the evolution of severe structural and functional injury may be averted during ALI/ARDS. TNX-832 (formerly known as Sunol-cH36), directed against human TF, which can block the pathological complications of TF-dependent thrombus formation. The blockage by TNX-832 of initiating events in the extrinsic coagulation pathway may attenuate the effects on pro-inflammatory events in ALI/ARDS patients, thereby averting or decreasing disordered fibrin deposition and averting the evolution of severe structural and functional injury.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Suspected or proven bacterial infection
3. Receiving positive pressure ventilation through an endotracheal tube
4. Have ALI/ARDS, defined as having all of the following:

   * bilateral infiltrates consistent with pulmonary edema
   * Hypoxemia
   * no clinical evidence of left atrial hypertension
5. Provide signed informed consent

Exclusion Criteria:

1. Mechanically or chemically-induced ALI/ARDS (including burns, trauma, and near drowning)
2. End-stage lung disease
3. Decompensated congestive heart failure
4. Authorization to withdraw life support
5. Hemoglobin persistently <8.0 g/dL
6. Subjects who have any one of the following:

   * platelet count <50,000/mm^3
   * prolonged prothrombin time (PT)
   * prolonged activated partial thromboplastin time (aPTT)
   * having significant potential for disseminated intravascular coagulation (DIC)
7. Subjects who have two or more of the following:

   * prolonged aPTT
   * fibrinogen level below the lower limit of normal
   * presence of petechiae, ecchymoses, or other evidence of coagulopathy
8. Subjects who have a history of one or more of the following:

   * hematuria (microscopic or gross)
   * urinary tract neoplasia
   * nephrolithiasis
   * glomerulonephritis
   * active urinary tract infection (UTI)
9. Bleeding disorders within the past 6 weeks or vasculitis with diffused alveolar hemorrhage
10. Diagnosis of bleeding peptic ulcer disease within the previous 2 months
11. Congenital bleeding diatheses such as hemophilia
12. Treatment with anti-platelet, anti-coagulant agents, or non-steroidal anti-inflammatory drugs (NSAIDs)within 72 hours following infusion of study drug

    * Therapeutic heparin:

      * Unfractionated heparin within eight hours prior to study drug infusion
      * Low molecular weight heparins within the 12 hours prior to study drug infusion
    * Prophylactic heparin:

      * Unfractionated heparin >15,000 units/day
      * Low molecular weight heparins
    * Warfarin if used within 7 days prior to study drug infusion
    * Thrombolytic treatment within 3 days prior to study drug infusion
    * 8Glycoprotein IIb/IIIa antagonists within 7 days prior to study drug infusion
    * Aspirin or any aspirin containing compound within 3 days prior to study drug infusion
    * APC infusion within 72 hours prior to study drug infusion
13. Major trauma or trauma subjects at an increased risk of bleeding
14. History of severe head trauma that required hospitalization, intracranial surgery, or stroke or any history of intracerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass lesion with an epidural catheter or who anticipate receiving an epidural catheter during study drug infusion
15. Major surgery within the previous 3 days, any postoperative subject with evidence of active bleeding, or any subject with planned or anticipated surgery within 72 hours after study drug infusion. History of abnormal bleeding during surgical procedures
16. Chronic renal failure, defined as a calculated glomerular filtration rate (GFR) ≤20 mL/min
17. Subjects with baseline aspartate transaminase (AST) or alanine transaminase (ALT) level >5 times the upper limit of normal. Subjects with known esophageal varices, chronic jaundice, biopsy proven cirrhosis, or chronic ascites
18. History of organ transplant (including bone marrow)
19. Subjects with malignancy having a life expectancy <6 months
20. Known human immunodeficiency virus (HIV) positive with CD4+ T Cell count <200/uL
21. Women who are pregnant or nursing
22. Participation in another clinical research study within 30 days before administration of study drug, with the exception of participation in studies involving noninvasive monitoring medical devices
23. Any prior treatment with a murine or chimeric antibody
24. Subjects who are moribund and where death is perceived to be imminent (within 72 hours after screening)
25. Subjects who have persistent hypotension not responding to fluid or vasopressor administration; subjects who require more than two vasopressors 26. Any medical condition which in the opinion of the investigator would interfere with optimal participation in the study or that would produce a significant risk to a subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hing Wong, PhD, Study Director — Altor BioScience
Locations (7):
- United States (6):
  - University of Miami, Miami, Florida
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Baylor School of Medicine, Houston, Texas
- Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Morris PE, Steingrub JS, Huang BY, Tang S, Liu PM, Rhode PR, Wong HC. A phase I study evaluating the pharmacokinetics, safety and tolerability of an antibody-based tissue factor antagonist in subjects with acute lung injury or acute respiratory distress syndrome. BMC Pulm Med. 2012 Feb 16;12:5. doi: 10.1186/1471-2466-12-5. PMID 22340260
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22340260/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; 0.06 MG/KG Dose; 0.1 MG/KG Dose; 0.08 MG/KG Dose: TNX-832
Period: Overall Study
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Started | 3 | 5 | 5 | 5
Completed | 3 | 5 | 4 | 4
Not Completed | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose | Total
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.67 (24.3) | 40.40 (18.2) | 54.60 (13.7) | 54.00 (16.9) | 49.53 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 3 | 14
  Male | 1 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 2 | 5
  White | 1 | 4 | 3 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Subjects with Acute Lung Injury/Acute Respiratory Distress Syndrome [Count of Participants; unit: Participants] | 3 | 5 | 5 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: To evaluate the safety of escalating dose levels of TNX-832 in subjects with suspected or proven bacteria-induced ALI/ARDS. Safety was assessed by number of treatment emergent adverse events, and changes in vital signs, ECGs, laboratory, coagulation and pulmonary function parameters from baseline. Immunogenicity (serum anti-TNX-832 antibody response) was evalutated.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 3 | 5 | 5 | 5
Participants | 3 | 4 | 5 | 4

2. Primary Outcome: Cmax
Description: maximum observed concentration (Cmax)
Time Frame: predose; 15 and 30 min; 1, 4, 6, 12 and 24 hrs; 2, 3, 4, 5, 6, and 7 days, 2, 3, 4 weeks
Population: O participants were analyzed for placebo pk
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 0 | 5 | 5 | 5
ng/mL |  | 1297 (560) | 1800 (253) | 1492 (344)

3. Primary Outcome: AUCinf and AUClast
Description: Area under the plasma concentration curve from time 0 extrapolated to infinite time (AUC0-inf).
  AUClast (area under the serum concentration-time curve from the time of dosing to the time of the last observed concentration).
Time Frame: Up 163.3 hours
Population: 0 participants were analyzed in the placebo AUCinf. Two participants in the 0.06 mg/kg and 1participant in the 0.1 mg/kg cohort did not meet the criteria for reliable estimation of PK parameters and are not included in calculation of Cohort mean values.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 0 | 3 | 4 | 5
mcg*hr/mL
  AUCinf |  | 39031 (24178) | 59921 (16629) | 59851 (20459)
  AUClast |  | 35868 (22950) | 53973 (17289) | 56860 (21705)

4. Primary Outcome: Terminal t1/2 and Tmax
Description: t1/2 (terminal elimination phase half life). Tmax (time to maximum serum concentration).
Time Frame: predose; 15 and 30 min; 1, 4, 6, 12 and 24 hrs; 2, 3, 4, 5, 6, and 7 days, 2, 3, 4 weeks
Population: 0 participants were analyzed in placebo Terminal t1/2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 0 | 3 | 4 | 5
hr
  T1/2 |  | 18.5 (5.9) | 22.6 (6.2) | 22.6 (3.1)
  Tmax |  | 1.0 (0.0) | 0.9 (0.4) | 4.2 (0.6)

5. Primary Outcome: Vd and Vss
Description: Volume of distribution (Vd) based on the terminal elimination phase, also referred to as VZ; in mL/kg.
  Volume of distribution at steady state (Vss), calculated as the Mean residence Time times Clearance; in mL/kg.
Time Frame: predose; 15 and 30 min; 1, 4, 6, 12 and 24 hrs; 2, 3, 4, 5, 6, and 7 days, 2, 3, 4 weeks
Population: 0 participants were analyzed in placebo Vd and Vss
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 0 | 3 | 4 | 5
mL/kg
  Vd |  | 46.1 (13.1) | 54.5 (6.6) | 47.7 (16.0)
  Vss |  | 44.9 (12.29) | 53.0 (5.3) | 46.7 (14.7)

6. Primary Outcome: Cl
Description: Total body clearance, CL=Dose/AUC; in mL/hr/kg
Time Frame: up to 1 week
Population: 0 participants were analyzed in placebo Cl
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
Number analyzed (Participants) | 0 | 3 | 4 | 5
mL/hr/kg |  | 1.9 (1.0) | 1.8 (0.4) | 1.5 (0.7)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Placebo | 0.06 MG/KG Dose | 0.1 MG/KG Dose | 0.08 MG/KG Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/5 | 2/5 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 4/5 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | 0.06 MG/KG Dose (N=5) | 0.1 MG/KG Dose (N=5) | 0.08 MG/KG Dose (N=5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
acute renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | 0.06 MG/KG Dose (N=5) | 0.1 MG/KG Dose (N=5) | 0.08 MG/KG Dose (N=5)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2
Lymphocytic infiltration (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Macroglossia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bloody discharge (General disorders) | 0 | 0 | 1 | 0
Edema peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 0 | 0
Candiduria (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Hematocrit decreased (Investigations) | 0 | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 5 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-02-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT01438853/Prot_SAP_000.pdf